CLINICAL TRIAL: NCT01427049
Title: The Evaluation of Renal Denervation on Several Biological Variables in Patients With Uncontrolled Hypertension. An Observational Feasibility Study.
Brief Title: The Effect of Renal Denervation on Biological Variables
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, P. J. Blankestijn, Dr, UMC Utrecht
Other Study IDs: 11-189; NL35945.041.11 (Other: CCMO)
Record Dates: First submitted 2011-08-16; First posted 2011-09-01 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Hypertension
Keywords: renal denervation; renal sympathetic denervation; renal ablation; resistant hypertension; hypertension; renal oxygenation; renal perfusion
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- renal denervation: Adults with a systolic BP ≥160 mmHg (≥150 mmHg for type 2 diabetics) with a stable drug regimen including 3 or more antihypertensive medications, including a diuretic, or inability to follow a stable drug regimen due to unacceptable side-effects of antihypertensive medication.
  Interventions: Device: renal denervation

INTERVENTIONS:
Device: renal denervation — percutaneous selective renal sympathetic denervation with the use of the Symplicity Catheter system
  Other Names: Symplicity Catheter system

SUMMARY:
Hypertension is a major and growing public health concern. Chronic elevation of sympathetic nervous system (SNS) activity has been identified as a major contributor to the complex pathophysiology of (essential) hypertension. The renal sympathetic nerves play a major role in the elevation of the SNS activity. Therapeutic renal denervation (RD), the deliberate disruption of the nerves connecting the kidneys with the central nervous system, has been shown to be an effective means of modulating elevated SNS activity - both by reducing the sympathetic modulation of renal function (renin release, sodium excretion and renal blood flow) and by removing the renal afferent sympathetic contribution to central blood pressure elevation.

This current study is an observational exploratory study. The main objective of this study is to learn more on the effects of RD. We wish to do that by quantifying the effects of RD on various biological variables. Those variables are studied in four sets of investigations: a radiological set, a laboratorial set, a set of blood pressure measurements and a set of investigations in the vascular laboratory. The radiological set consists of imaging of the heart and kidney function (renal perfusion) and structure (renal arteries), the laboratorial set of serum and urine tests, 24 h- home- and office- blood pressure measurements will be taken and finally the set of vascular tests contains investigations on pulse wave velocity(PWV) and heart rate variability(HRV). The data will most likely help us to define future studies, to describe the mode of action and the effects of RD on various organs and systems in more detail, and finally to define in more detail which type of hypertensive patients is especially likely to benefit of the procedure.

Hypothesis:

* We hypothesize that LV mass will decrease after RD. Because all patients have severe hypertension, it is likely that a substantial percentage will have increased LV mass.
* We hypothesize that renal perfusion and renal oxygenation increase after RD.
* We hypothesize that there will be no complications related to the device or procedure.
* We hypothesize that renal denervation has a beneficial effect on insulin resistance
* We hypothesize that renal denervation will decrease the blood pressure(office and 24-hour-measurements)
* We hypothesize that RD has a beneficial effect on PWV and HRV.

DETAILED DESCRIPTION:
Objective: The objectives of this study are: the investigation of changes in left ventricular mass (LV mass) after RD using MRI, renal perfusion and renal oxygenation after RD using dynamic contrast enhanced MRI (DCE MRI)and blood oxygenation level dependent MRI (BOLD MRI), the evaluation of safety of RD, in terms of structural changes in the renal arteries and kidney using Magnetic resonance angiography (MRA). Secondly the evaluation of changes in various biological functions assessed by analysis of blood and/or urine samples. Thirdly the quantification of changes in blood pressure. Finally the changes in pulse wave velocity (PWV) and heart rate variability (HRV).

Study design: Observational exploratory-study.

Study population: Adults with a systolic BP ≥160 mmHg (≥150 mmHg for type 2 diabetics) with a stable drug regimen including 3 or more antihypertensive medications, including a diuretic, or inability to follow a stable drug regimen due to unacceptable side-effects of antihypertensive medication.

Main study parameters/endpoints: The effect of RD on: radiological variables: left ventricular wall mass, renal perfusion, renal oxygenation and the anatomy of the renal arteries. Secondly the effect of RD on biological variables assessed by analysis of blood and/or urine samples. Thirdly the changes in blood pressure. Finally the changes in PWV and HRV after RD.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The risks associated with the tests and procedures performed for the clinical study are limited. There are no known risks associated with MRI when appropriate safety guidelines are followed. Based on the experience form our previous studies, we do not expect any potential risks regarding the cessation of anti-hypertensives.

ELIGIBILITY:
Inclusion Criteria:

* Individual has a systolic BP ≥160 mmHg (≥150 mmHg for type 2 diabetics) based on an average of 3 office BP readings measured according to the guidelines in appendix A.
* Individual is adhering to a stable drug regimen including 3 or more antihypertensive medications, including a diuretic (with no changes for a minimum of 2 weeks prior to enrolment) which is expected to be maintained for at least 6 months. Or:
* Has experienced side effects to several anti-hypertensive medications
* Individual is ≥18 years of age.
* Individual agrees to have all study procedures performed, and is competent and willing to provide written, informed consent to participate in this clinical study.

Exclusion Criteria:

* Individual has a treatable secondary cause of hypertension. (it is possible that during baseline procedures secondary causes of hypertension are discovered, those individuals will be excluded from participation of the study.)
* Individual has renal artery anatomy that is ineligible for treatment including:
* Main renal arteries < 4 mm in diameter or < 20 mm in length.
* Hemodynamically or anatomically significant renal artery abnormality or stenosis in either renal artery which, in the eyes of the operator, would interfere with safe cannulation of the renal artery or meets standards for surgical repair or interventional dilation.
* A history of prior renal artery stenting.
* Multiple main renal arteries in either kidney.
* Individual has an estimated glomerular filtration rate (eGFR) of <30mL/min/1.73m2, using the MDRD calculation.
* Individual has type 1 diabetes mellitus.
* Individual has experienced a myocardial infarction, unstable angina pectoris, or a cerebrovascular accident within 6 months of the screening visit, or has widespread atherosclerosis, with documented intravascular thrombosis or unstable plaques.
* Individual has scheduled or planned surgery or cardiovascular intervention in the next 6 months.
* Individual has hemodynamically significant valvular heart disease for which reduction of BP would be considered hazardous.
* Individual has an implantable cardioverter defibrillator (ICD) or pacemaker whose settings cannot allow for RF energy delivery.
* Individual has any serious medical condition, which in the opinion of the investigator, may adversely affect the safety and/or effectiveness of the participant or the study (i.e., patients with clinically significant peripheral vascular disease, abdominal aortic aneurysm, bleeding disorders such as thrombocytopenia, haemophilia, or significant anaemia, or arrhythmias such as atrial fibrillation).
* Individual is pregnant, nursing or planning to be pregnant.
* Individual has a known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or would be unlikely or unable to comply with study follow-up requirements.
* Individual is currently enrolled in another investigational drug or device trial.
* Individual is currently being treated with any of the following medications:

  1. Drugs that cause salt retention (e.g., systemic corticosteroids and fludrocortisone)
  2. Warfarin or phenprocoumon that cannot be temporarily stopped for the procedure.
* Any contraindications for MRI:

  1. The presence of implanted cardiac pacemakers and/or auto-implanted cardioverter defibrillators.
  2. Mechanical cardiac valves.
  3. Implanted electronic devices like cochlear implants and nerve stimulators.
  4. Patients who are unable to fit into the bore of the magnet.
  5. Claustrophobia.
  6. Prosthesis of a joint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a systolic BP ≥160 mmHg (≥150 mmHg for type 2 diabetics) with a stable drug regimen including 3 or more antihypertensive medications, including a diuretic, or inability to follow a stable drug regimen due to unacceptable side-effects of antihypertensive medication.
  This current study is an observational exploratory-study.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2011-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in Blood pressure related endpoints: | t=0, t=6 and t=12 months
  * Incidence of achieving target systolic blood pressure(SBP) (SBP <140 mmHg, or <130 for diabetics)
  * Incidence of achieving a >10 mmHg reduction in SBP
  * Change in office BP from baseline to 6 months post-renal denervation.
  * Change in 24 hour ambulatory blood pressure taken without the use of antihypertensive medication, from baseline to 12 months post-renal denervation.
  * Changes in SBP and diastolic blood pressure (DBP) from baseline to 6 and 12 months

SECONDARY OUTCOMES:
Radiologic endpoint | t=0 and t=12 months
  - The change in left ventricular mass -determined by balanced SSFP cine MRI - after renal denervation compared with baseline. This change will be expressed in grams and grams per square meter of body surface area.
radiologic endpoint | t=0 and t=12 months
  The change of renal perfusion 12 months after renal denervation compared to baseline. Dynamic contrast-enhanced MRI will be used for quantitative assessment of renal perfusion. Renal perfusion will be calculated in mL/gram/min.
radiologic endpoint | t=0 and t=12 months
  The change of renal oxygenation after renal denervation compared to baseline; Changes in oxygenation are calculated in changes in T2 * ratio (i.e. T2 * cortex/ T2 * medulla).
radiologic endpoint | t=0 and t=12 months
  - the change in the anatomy of the renal arteries 12 months after renal denervation compared to baseline. for example the existing of renal artery stenosis 12 months after renal denervation compared to baseline: New renal artery stenosis > 60% confirmed by angiogram.
laboratorial endpoint | t=0 and t=12 months
  Absolute changes of: eGFR, plasma renin activity (PRA), aldosterone, ACE, lipid spectrum, proteinuria, insulin, C-peptide, glucose, VMA, metanephrines and catecholamines, 12 months after renal denervation compared to baseline measurements
blood pressure related endpoint | t=0 t=6 and t=12 months
  The effect of renal denervation on the development of orthostatic hypotension
  - The change in the existing of orthostatic hypotension at baseline compared with the existing at 6 and 12 months after renal denervation will be determined
blood pressure related endpoint | t=0 and t=12 months
  The change in the effect of blood pressure, renin and aldosterone in the captopril test 12 months after renal denervation compared with the baseline measurements:
  Change in blood pressure reaction on captopril. Change in the effect of captopril on absolute changes of aldosterone and renin.
blood pressure related endpoint | measured every month after renal denervation
  The change in home blood pressure measurements during 12 months after renal denervation
endpoint derived from investigations at the vascular laboratory | t=0 and t=12 months
  The in heart rate variability 12 months after renal denervation compared with the baseline measurement
  Change in LF/HF-ratio. Change in LF-power.
endpoint derived from investigations at the vascular laboratory | t=0 and t=12 months
  The change of pulse wave velocity 12 months after renal denervation compared with the baseline measurement:
  Change in peripheral pressure pulse waveform. Change in central aortic pressure waveform. Change in Augmentation Index (AI).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Blankestijn, Dr., Principal Investigator — UMC Utrecht department of Nephrology and Hypertension; Eva Vink, PhD Student, Principal Investigator — UMC Utrecht Department of Nephrology and Hypertension
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Blankestijn PJ, Ritz E. Renal denervation: potential impact on hypertension in kidney disease? Nephrol Dial Transplant. 2011 Sep;26(9):2732-4. doi: 10.1093/ndt/gfr190. Epub 2011 Apr 19. No abstract available. PMID 21505095
- [Background] Symplicity HTN-2 Investigators; Esler MD, Krum H, Sobotka PA, Schlaich MP, Schmieder RE, Bohm M. Renal sympathetic denervation in patients with treatment-resistant hypertension (The Symplicity HTN-2 Trial): a randomised controlled trial. Lancet. 2010 Dec 4;376(9756):1903-9. doi: 10.1016/S0140-6736(10)62039-9. Epub 2010 Nov 17. PMID 21093036
- [Background] Symplicity HTN-1 Investigators. Catheter-based renal sympathetic denervation for resistant hypertension: durability of blood pressure reduction out to 24 months. Hypertension. 2011 May;57(5):911-7. doi: 10.1161/HYPERTENSIONAHA.110.163014. Epub 2011 Mar 14. PMID 21403086
- [Background] Siddiqi L, Joles JA, Grassi G, Blankestijn PJ. Is kidney ischemia the central mechanism in parallel activation of the renin and sympathetic system? J Hypertens. 2009 Jul;27(7):1341-9. doi: 10.1097/HJH.0b013e32832b521b. PMID 19444143
- [Background] Krum H, Schlaich M, Whitbourn R, Sobotka PA, Sadowski J, Bartus K, Kapelak B, Walton A, Sievert H, Thambar S, Abraham WT, Esler M. Catheter-based renal sympathetic denervation for resistant hypertension: a multicentre safety and proof-of-principle cohort study. Lancet. 2009 Apr 11;373(9671):1275-81. doi: 10.1016/S0140-6736(09)60566-3. Epub 2009 Mar 28. PMID 19332353
- [Derived] Verloop WL, Vink EE, Spiering W, Blankestijn PJ, Doevendans PA, Bots ML, Vonken EJ, Voskuil M, Leiner T. Effects of renal denervation on end organ damage in hypertensive patients. Eur J Prev Cardiol. 2015 May;22(5):558-67. doi: 10.1177/2047487314556003. Epub 2014 Oct 17. PMID 25326543